CLINICAL TRIAL: NCT02397174
Title: Mediterranean Diet Versus Hypocaloric Diet: What is the Best Choice for the Treatment of Polycystic Ovary Syndrome (PCOS)?
Brief Title: Mediterranean Diet Versus Hypocaloric Diet in PCOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona (Other)
Collaborators: Federico II University (Other); University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Francesco Orio, prof, Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIEMED1
Record Dates: First submitted 2015-03-06; First posted 2015-03-24 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary syndrome; hypocaloric diet; Ovarian Cysts; Ovarian Diseases; Obesity; Mediterranean Diet
MeSH Terms: conditions — Polycystic Ovary Syndrome; Ovarian Cysts; Ovarian Diseases; Obesity | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mediterranean Diet (Experimental): The diet programme will be characterized by carbohydrates (60 %); proteins (20 %, half comprised of vegetable proteins); total fat (20 %; saturated fat < 10 %). After calculating the patient's energy need, the amount of calories will be successively adjusted to create an 800 kcal deficit per day.
  Interventions: Other: mediterranean diet, restricted calorie
- hypocaloric diet (Active Comparator): The diet programme will be characterized by carbohydrates (50%),total lipids (30%) and proteins (20%). After calculating the patient's energy need, the amount of calories will be successively adjusted to create an 800 kcal deficit per day.
  Interventions: Other: hypocaloric diet, restricted calorie

INTERVENTIONS:
Other: mediterranean diet, restricted calorie — 50 pcos women will be assigned to hypocaloric mediterranean diet for 6 months
  Arms: Mediterranean Diet
Other: hypocaloric diet, restricted calorie — 50 pcos women will be assigned to standardized hypocaloric diet for 6 months
  Arms: hypocaloric diet

SUMMARY:
Polycystic ovary syndrome (PCOS) is the most common endocrinopathy of reproductive-aged women that manifests itself with chronic anovulation, hyperandrogenism and insulin resistance. Available guidelines recommend lifestyle intervention although they do not suggest the best dietetic regimen for the treatment of PCOS. Thus, the purpose of this study is to compare the effectiveness of two nutritional protocols, namely Mediterranean Diet and Hypocaloric Diet in PCOS women.

DETAILED DESCRIPTION:
PCOS is the most common endocrine disorder of reproductive age women, that is often associated with chronic anovulation, hyperandrogenism and insulin resistance. The central importance of insulin resistance in the pathogenesis of the syndrome has been established by several in vivo and in vitro studies. No data are available for the best therapeutical approach for metabolic dysfunction of PCOS. The new guidelines for the management of metabolic risk in PCOS strongly recommended that overweight/obese women with PCOS should lose weight changing their lifestyle. Although calorie-restricted diets are currently recommended to reach the healthy weight, there are still unsatisfied data regarding the best dietetic regimen that should be suggested.

In this study, our purpose is to compare two nutritional protocols in order to find the best dietetic approach for improving clinical, metabolic and hormonal outcomes in pcos women.

ELIGIBILITY:
Inclusion Criteria:

* Polycystic ovary syndrome (using ESHRE/ARSM 2007 criteria)
* BMI > 25

Exclusion Criteria:

* Age <18 or >35 years
* BMI higher than 35
* Pregnancy
* Hypothyroidism, hyperprolactinemia, Cushing's syndrome, nonclassical congenital adrenal hyperplasia, use of oral contraceptives, glucocorticoids, antiandrogens, ovulation induction agents, antidiabetic or antiobesity drugs or other hormonal drugs within the previous 6 months
* Subjects with neoplastic, metabolic (including glucose intolerance), hepatic, and cardiovascular disorder or other concurrent medical illness (i.e. diabetes, renal disease, or malabsorptive disorders, cephalea)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
improvement in insulin resistance measured by HOMA index | 6 months

SECONDARY OUTCOMES:
composite improvement in clinical parameters (Body mass index, normalization of menses, hirsutism, waist to hip ratio); | 6 months
composite improvement in metabolic parameters (total, LDL and HDL cholesterol); | 6 months
composite improvement in hormonal parameters (Testosterone, Androstenedione, DHEAS, FSH, LH, beta estradiol) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Orio, MD, Principal Investigator — Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona
Locations (1):
- Fertility Techniques SSD,Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona, Salerno, Salerno, Italy

REFERENCES:
- [Result] Palomba S, Giallauria F, Falbo A, Russo T, Oppedisano R, Tolino A, Colao A, Vigorito C, Zullo F, Orio F. Structured exercise training programme versus hypocaloric hyperproteic diet in obese polycystic ovary syndrome patients with anovulatory infertility: a 24-week pilot study. Hum Reprod. 2008 Mar;23(3):642-50. doi: 10.1093/humrep/dem391. Epub 2007 Dec 23. PMID 18158291
- [Result] Palomba S, Falbo A, Giallauria F, Russo T, Rocca M, Tolino A, Zullo F, Orio F. Six weeks of structured exercise training and hypocaloric diet increases the probability of ovulation after clomiphene citrate in overweight and obese patients with polycystic ovary syndrome: a randomized controlled trial. Hum Reprod. 2010 Nov;25(11):2783-91. doi: 10.1093/humrep/deq254. Epub 2010 Sep 21. PMID 20858697